CLINICAL TRIAL: NCT00166595
Title: Pharmacogenetics of Risperidone in Children With Pervasive Developmental Disorder (PDD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: PPRU 10545s
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2012-07

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Risperidone; Autism; Pervasive Developmental Disorder (PDD)
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to determine if the known differences in genes influence drug metabolizing enzymes and receptors that are involved in risperidone drug action. The study will determine if differences in these genes will change the concentration of risperidone in the blood over time in children in relation to side effects and clinical response to risperidone.

DETAILED DESCRIPTION:
To the knowledge of the investigators there are no studies documenting the pharmacokinetics and pharmacogenetics of risperidone in children with PDD. Currently the PPRU network is conducting a PK study whose aim is to establish a new enantio-selective micro-assay methodology and to generate preliminary population PK data of risperidone and its metabolites in PDD. This study focuses on pharmacogenetic evaluation of PDD patients having little or no effect, those that are unusually sensitive and those experiencing drug toxicity/adverse events at standard risperidone dosages.

In this study two 5 ml blood samples will be drawn at a regulary scheduled PK visit. Alternatively pooled waste blood samples or a buccal swab can be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 4 and 21 years.
* Patients meeting DSM-IV criteria for autistic disorder, Pervasive Developmental Disorder (PDD), or Pervasive Developmental Disorder-Not Otherwise Specified (PDD-NOS) and about to initiate clinical treatment or currently clinically treated with risperidone.
* Patients about to initiate clinical treatment or currently clinically treated with risperidone, or currently on risperidone as a participant in one of the multi-site Research Unit for Pediatric Psychopharmacology (RUPP) protocols.

Exclusion Criteria:

* Children taking psychotropic or other medication that will significantly interact with target CYP 450 isoenzyme activity, such to the discretion of the principal investigator (PI).
* Patients with known renal or hepatic dysfunction (e.g. serum creatinine, and transaminases or bilirubin exceeding age specific upper range limits) are not eligible.
* Failure of the parent/legal guardian to give informed consent.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 2003-02; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospital of Michigan/Wayne State University, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio